CLINICAL TRIAL: NCT04986514
Title: Identification of Biomarkers Associated With Disease Worsening Within 10 Years in Scleroderma Patients
Brief Title: Implementation of a Biological Sample Collection in Systemic Sclerosis Patients
Acronym: SCLERO-BIOBANK
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_58; 2021-A00107-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-04

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Biomarkers; Bio-banking
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum (3 aliquots) and plasma (3 aliquots)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with systemic sclerosis
  Interventions: Other: Bio-banking without genetic analysis

INTERVENTIONS:
Other: Bio-banking without genetic analysis — For patients included in SCLERO-BIOBANK study, 2 blood samples will be collected at each SSc evaluation (usually once a year), in addition to the routine care blood collection.

SUMMARY:
Systemic sclerosis (SSc) is the most severe of the systemic autoimmune diseases. It is characterized by skin and organ fibrosis (mainly interstitial lung disease, which affects 40-50% of patients), as well as severe vascular complications such as pulmonary hypertension (5-10%), renal crisis (2%), and digital gangrene (5%). There are currently no validated prognostic biomarkers for the progression of SSc, yet it is crucial to better predict the progression of SSc to optimize patient management, but also to identify the optimal population for clinical trials ("progressor" patients). Furthermore, there are no validated biomarkers of response to immunosuppressive therapies that would be useful both in patient management and in the evaluation of new treatments in clinical trials. The internal medicine department of the Lille University Hospital is a national and European reference center for the management of patients with SSc. Nearly 500 patients are followed annually in the internal medicine department. As part of their routine care, patients are hospitalized in average once a year in the internal medicine department of the Lille University Hospital for a complete assessment of their SSc. This assessment includes a detailed medical observation, complementary examinations and blood and urine biology tests. The purpose of this study would be to collect 2 additional blood samples during the standard evaluation of scleroderma patients. The main objective of this collection of biological samples for scientific research will be the identification of new biomarkers associated with prognosis and treatment response to improve the management of SSc patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed for SSc in the internal medicine or cardiology department of the Lille University Hospital
* Fulfilling the ACR/EULAR and/or VEDOSS criteria for SSc
* Being insured by the French social security system
* Having the ability to understand the requirements of the study and provide informed consent

Exclusion Criteria:

* Administrative reasons: unable to receive informed information, lack of social security coverage
* Pregnant or lactating women
* Persons deprived of liberty
* Minors or protected adults
* Persons who have refused or are unable to give informed consent
* Persons in emergency situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient followed for SSc in the internal medicine or cardiology department of the Lille University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2043-04 (Estimated); Study Completion 2043-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence during the follow-up period of an aggravation defined as death, onset or worsening of organ damage | Through study completion an average of 10 years
  Identify biomarkers that are associated with disease prognosis and treatment response during 10 years of follow-up.

SECONDARY OUTCOMES:
EUSTAR score | Baseline and through study completion, an average of 10 years
  Identify new biomarkers associated with disease severity and disease activity at study entry and the evolution of disease severity and activity over time
Medsger score | Baseline and through study completion, an average of 10 years
  Identify new biomarkers associated with disease severity and disease activity at study entry and the evolution of disease severity and activity over time

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille